CLINICAL TRIAL: NCT05621512
Title: Workplace Intervention Among Pregnant Hospital Employees - a Cluster Randomized Trial
Brief Title: Workplace Intervention Among Pregnant Hospital Employees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region MidtJylland Denmark (Other)
Collaborators: Defactum, Central Denmark Region (Other Government); Aarhus University Hospital (Other); Herning Hospital (Other)
Responsible Party: Principal Investigator, Rikke Damkjær Maimburg, Ass. prof., University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29-2019-03
Record Dates: First submitted 2022-06-16; First posted 2022-11-18 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Sick Leave; Pregnancy; Midwifery
Keywords: Risk factors; Health Care Professionals; Intervention; Workplace

STUDY DESIGN:
Intervention Model Description: Cluster randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention implies a letter of invitation for a session between the employee, the department manager, and a midwife concerning workplace risk assessment and agreement on feasible work adjustments if necessary. A second session within gestational week 26-28 is scheduled to follow-up and readjust if necessary. A systematic frame for sessions is developed by the research team and conclusions from the sessions are registered within a piloted standardized template.
  The employee and the manager can initiate contact with the midwife at any time, e.g in case of new symptoms or discomfort and need for support or guidance. If sick leave is considered, a new session is recommended and may be scheduled at any time.
  To ensure transparency of guidance and workplace adjustments for other relevant healthcare professionals, the employee is asked to inform her general practitioner (GP) and midwife of the program.
  Interventions: Other: Preventive sessions
- Usual practice (No Intervention): Hospital pregnancy policy is usual practice and implies a meeting between the pregnant employee and her manager concerning an individual risk assessment. A risk assessment-template can be downloaded from the hospital website.
  If minimizing potential risks by adjustments is not possible the employee should be redeployed. If redeployment is not possible the pregnant employee may be absent due to pregnancy related symptoms.
  The pregnant employee is requested to inform her GP about agreements.

INTERVENTIONS:
Other: Preventive sessions — Preventive sessions between the pregnant employee, her manager and a midwife.
  Arms: Intervention

SUMMARY:
The aim of this study is to reduce sick leave and improve wellbeing. This is measured as physical and mental health, general work ability, work-life balance, manager support and completed work adjustments among pregnant health care professionals. It is hypothesised that pregnant employees participating in preventive sessions with their manager and a midwife in addition to the hospital standard pregnancy policy management will have less sick leave and report better wellbeing compared to the reference group.

DETAILED DESCRIPTION:
Sick leave during pregnancy is frequent and studies report proportions of employees on sick leave between 36-75%. Reasons for sick leave in early pregnancy are nausea, vomiting and dizziness whereas Braxton Hicks contractions, low back and pelvic girdle pain are more common in late pregnancy. Further, sick leave is strongly associated with working conditions and appropriate work adjustment.

The study design is cluster randomization with participation of all departments at Aarhus University Hospital (AUH), Denmark. Half of the departments are randomized to the intervention and the remaining to the reference group. The intervention group will receive a protocolized intervention with midwifery support as an add-on to usual practice. The reference group will receive protocolized usual practice.

Data are obtained from the hospital payment system and by survey (RedCap).

The sample size is calculated to find a difference of ≥ 7 days with a standard deviation of 25. To achieve a statistical power of 80% with a significance level of p ≤ 0.05 an estimated 202 participants will be required in each of the groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant employees working as health care professionals at Aarhus University Hospital

Exclusion Criteria:

* Gest. week > 20

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 404 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of days on sick leave | gestational period until gestational week 32
  Sick leave is specified by mean number of days on sick leave and the proportion of employees on sick leave throughout pregnancy and within trimesters (first trimester defined as gestational week 1 - 12, second trimester being gestational week 13 - 27 and third trimester being gestational week 28 - maternity leave)

SECONDARY OUTCOMES:
Self-rated health | at inclusion and at gestational week 30
  Self-rated health is explored with the item from Short Form 36 Health Survey Questionnaire: "In general, would you say your health is?: Excellent, very good, good, fair and poor?" Item values are coded from 1-5 with 1 being "excellent". Self-rated health is specified by mean scores.
Work ability | At inclusion and at gestational week 30
  Work ability is explored with three items from The Work Ability Index: "Assume that your work ability at its best has a value of 10 points. How many points would you give to your current work ability?" with answers on a scale from 1-10. Furthermore, "How do you rate your current work ability with respect to the physical demands of your work?" and "How do you rate your current work ability with respect to the mental demands of your work?" are included with response choices: "Very good, rather good, moderate, rather poor, very poor". Answers are coded 1-5 with 1 being "very poor". Work ability is specified by mean scores.
Psycho-social working environment | At inclusion and at gestational week 30
  The Copenhagen Psychosocial Questionnaire short version (COPSOQ) explores psycho-social working environment with the items: "How often have you felt worn out?" and "How often have you been emotionally exhausted?". Response choices are: "All the time, a large part of the time, part of the time, a small part of the time, not at all". Responses are coded from 1-5 with 1 being "all the time". The dimension of influence is explored with the questions: "Do you have a large degree of influence concerning your work?" and "Can you influence the amount of work assigned to you?" with response choices: "Always, often, sometimes, seldom, never/hardly ever". Answers are coded 1-5 with 1 being never/hardly. Psycho-social working environment is specified by mean scores.
Relation to immediate superior | At inclusion and at gestational week 30
  COPSOQ explores the dimension of relation to immediate superior is included with the items: "To what extend would you say that your immediate superior gives high priority to job satisfaction?" and "To what extend would you say that your immediate superior is good at work planning" Response choices are: "To a very large extend, to a large extend, somewhat, to a small extend, to a very small extend". Answers are coded from 1-5 with 1 being "to a very small extend". Relation to immediate superior is specified by mean scores.
Influence | At inclusion and at gestational week 30
  COPSOQ explores the dimension of influence is explored with the questions: "Do you have a large degree of influence concerning your work?" and "Can you influence the amount of work assigned to you?" with response choices: "Always, often, sometimes, seldom, never/hardly ever". Answers are coded 1-5 with 1 being never/hardly. Influence is specified by mean scores.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Maribo, Reseracher, Study Chair — Region MidtJylland Denmark
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided